CLINICAL TRIAL: NCT04466007
Title: Multicenter, Randomized, Dose-search, Parallel, Double-blind, and Placebo-controlled Clinical Trial to Evaluate the Safety and Efficacy of Intramuscular Administration of Allogeneic Adipose Tissue Adult Mesenchymal Stem Cells in Diabetic Patients With Critical Limb Ischemia Without Possibility of Revascularization
Brief Title: Safety and Efficacy of Allogeneic Adipose Tissue Mesenchymal Stem Cells in Diabetic Patients With Critical Limb Ischemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Collaborators: Clinica Universidad de Navarra, Universidad de Navarra (Other); Hospital Universitario La Paz (Other); Gregorio Marañón Hospital (Other); Hospital Clínico Universitario de Valladolid (Other); Hospital Universitario Virgen de la Arrixaca (Other); University of Salamanca (Other); Hospital General Universitario de Alicante (Other); Hospital Universitario La Fe (Other); Hospital Victoria Eugenia Cruz Roja Española (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NOMA (No More Amputations)
Record Dates: First submitted 2020-07-01; First posted 2020-07-10 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2024-10

CONDITIONS: Limb Ischemia; Diabetic Foot
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control arm (Placebo Comparator): 0.9% physiological saline
  Interventions: Drug: Placebos
- Low dose treatment arm (Experimental): Low dose allogeneic mesenchymal stem cells derived from adipose tissue
  Interventions: Drug: Low dose allogeneic mesenchymal stromal cells
- High dose treatment arm (Experimental): High dose allogeneic mesenchymal stem cells derived from adipose tissue
  Interventions: Drug: High dose allogeneic mesenchymal stromal cells

INTERVENTIONS:
Drug: High dose allogeneic mesenchymal stromal cells — Allogeneic mesenchymal stromal cells derived from adipose tissue administered intramuscularly
  Arms: High dose treatment arm
Drug: Low dose allogeneic mesenchymal stromal cells — Allogeneic mesenchymal stromal cells derived from adipose tissue administered intramuscularly
  Arms: Low dose treatment arm
Drug: Placebos — 0,9% physiological saline
  Arms: Control arm

SUMMARY:
Phase II national, multicenter, double-blind, randomized, placebo-controlled, phase-3 clinical trial of 3 parallel groups.

DETAILED DESCRIPTION:
Disease or disorder under study: Critical ischemia of the lower limbs in diabetic patients without the possibility of revascularization.

Main valuation variable: Proportion of Adverse Events related to treatment.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet ALL of the following criteria to be included in the study:

* Patients of both sexes.
* Age between 40 and 90 years.
* Severe grade vascular arteriosclerosis (category RB 4 and 5 mono or bilateral).
* Impossibility of surgical or endovascular revascularization or failure in revascularization surgery performed, at least 30 days before inclusion in the study, defining failure as direct non-arrival of vessels to the plantar arch.
* Normal biochemical parameters defined by:

  * Leukocytes> 3000 / mm3
  * Neutrophils> 1500 / mm3
  * Platelets> 100,000 / mm3
  * AST / ALT <2.5x upper limit of normal
* In patients with an ischemic ulcer, it must be stable for at least 1 week.
* Patients under conventional medical treatment for CLI.
* Women of childbearing age must obtain a negative result in a urine pregnancy test performed at the time of inclusion in the study and commit to using an effective contraceptive method during their participation in the study.
* Patients who have not participated in any other clinical trial during the 3 months prior to the inclusion visit.
* Patients who sign the informed consent.

Exclusion Criteria:

Patients who present SOME of the following criteria may not be selected to participate in this study:

* CLI with tissue loss in the target member (category 6 of RB).
* Previous major amputation in the target member.
* Uncontrolled hypertension (defined as PAS> 180 or PAD> 110 in at least 2 determinations during the selection period).
* Patients with severe heart failure or ejection fraction less than 30%.
* Patients with a previous diagnosis of ventricular arrhythmias or unstable angina.
* Patients with septicemia.
* Patients diagnosed with deep vein thrombosis in the 3 months prior to their inclusion in the study.
* Concomitant therapy that includes hyperbaric oxygen, angiogenic agents or Cox II inhibitors.
* Contraindication to perfusion NMR.
* Proliferative retinopathy without treatment.
* Diabetic nephropathy in hemodialysis.
* Patients previously treated with cell therapy, gene therapy or growth factors in the last year.
* Concomitant disease that limits life expectancy to 1 year or that does not ensure the follow-up period.
* Patients who have suffered a stroke or myocardial infarction in the 3 months prior to the inclusion visit.
* Severe anemia (hemoglobin <7.9g / dl) in the inclusion analysis.
* Patients with a previous diagnosis of chronic alcoholism.
* Any clinically significant anomaly detected in the Selection Period and which, in the opinion of the investigator, constitutes an impediment to the correct participation of the patient in the study or the fulfillment of the procedures established therein.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
Complication rate after treatment administration | 1 year

SECONDARY OUTCOMES:
Evaluation of vascularization though RMN | 1 year
Rutherford-Becker scale | 1 year
Wifi scale | 1 year
Ankle arm index | 1 year
Temperature | 1 year
  (ºC)
Twin perimeter | 1 year
  (cm)
Neuropathic symptoms (altered sensitivity) | 1 year
% amputations | 1 year

OTHER OUTCOMES:
SF-12 questionnaire | 1 year
VascuQol-6 questionnaire | 1 year

CONTACTS AND LOCATIONS:
Locations (10):
- Spain (10):
  - Hospital General de Alicante, Alicante
  - Hospital Gregorio Marañon, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - La Paz University Hospital, Madrid
  - Hospital Clinico Universitario Virgen de la Arrixaca, Murcia
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Victoria Eugenia Cruz Roja Española, Seville
  - Hospital Universitario La Fe, Valencia
  - Hospital de Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Garcia-Olmo D, Schwartz DA. Cumulative Evidence That Mesenchymal Stem Cells Promote Healing of Perianal Fistulas of Patients With Crohn's Disease--Going From Bench to Bedside. Gastroenterology. 2015 Oct;149(4):853-7. doi: 10.1053/j.gastro.2015.08.038. Epub 2015 Aug 24. No abstract available. PMID 26311275
- [Background] Garcia-Olmo D, Garcia-Arranz M, Herreros D, Pascual I, Peiro C, Rodriguez-Montes JA. A phase I clinical trial of the treatment of Crohn's fistula by adipose mesenchymal stem cell transplantation. Dis Colon Rectum. 2005 Jul;48(7):1416-23. doi: 10.1007/s10350-005-0052-6. PMID 15933795
- [Background] Garcia-Olmo D, Herreros D, Pascual I, Pascual JA, Del-Valle E, Zorrilla J, De-La-Quintana P, Garcia-Arranz M, Pascual M. Expanded adipose-derived stem cells for the treatment of complex perianal fistula: a phase II clinical trial. Dis Colon Rectum. 2009 Jan;52(1):79-86. doi: 10.1007/DCR.0b013e3181973487. PMID 19273960
- [Background] Panes J, Garcia-Olmo D, Van Assche G, Colombel JF, Reinisch W, Baumgart DC, Dignass A, Nachury M, Ferrante M, Kazemi-Shirazi L, Grimaud JC, de la Portilla F, Goldin E, Richard MP, Diez MC, Tagarro I, Leselbaum A, Danese S; ADMIRE CD Study Group Collaborators. Long-term Efficacy and Safety of Stem Cell Therapy (Cx601) for Complex Perianal Fistulas in Patients With Crohn's Disease. Gastroenterology. 2018 Apr;154(5):1334-1342.e4. doi: 10.1053/j.gastro.2017.12.020. Epub 2017 Dec 24. PMID 29277560
- [Background] Panes J, Garcia-Olmo D, Van Assche G, Colombel JF, Reinisch W, Baumgart DC, Dignass A, Nachury M, Ferrante M, Kazemi-Shirazi L, Grimaud JC, de la Portilla F, Goldin E, Richard MP, Leselbaum A, Danese S; ADMIRE CD Study Group Collaborators. Expanded allogeneic adipose-derived mesenchymal stem cells (Cx601) for complex perianal fistulas in Crohn's disease: a phase 3 randomised, double-blind controlled trial. Lancet. 2016 Sep 24;388(10051):1281-90. doi: 10.1016/S0140-6736(16)31203-X. Epub 2016 Jul 29. PMID 27477896
- [Background] Sanz-Baro R, Garcia-Arranz M, Guadalajara H, de la Quintana P, Herreros MD, Garcia-Olmo D. First-in-Human Case Study: Pregnancy in Women With Crohn's Perianal Fistula Treated With Adipose-Derived Stem Cells: A Safety Study. Stem Cells Transl Med. 2015 Jun;4(6):598-602. doi: 10.5966/sctm.2014-0255. Epub 2015 Apr 29. PMID 25925838
- [Background] Dormandy JA, Rutherford RB. Management of peripheral arterial disease (PAD). TASC Working Group. TransAtlantic Inter-Society Consensus (TASC). J Vasc Surg. 2000 Jan;31(1 Pt 2):S1-S296. No abstract available. PMID 10666287
- [Background] Gensler SW, Haimovici H, Hoffert P, Steinman C, Beneventano TC. Study of vascular lesions in diabetic, nondiabetic patients. Clinical, arteriographic, and surgical considerations. Arch Surg. 1965 Oct;91(4):617-22. doi: 10.1001/archsurg.1965.01320160071016. No abstract available. PMID 5836112
- [Background] Ciavarella A, Silletti A, Mustacchio A, Gargiulo M, Galaverni MC, Stella A, Vannini P. Angiographic evaluation of the anatomic pattern of arterial obstructions in diabetic patients with critical limb ischaemia. Diabete Metab. 1993 Nov-Dec;19(6):586-9. PMID 8026611
- [Background] Ouriel K. Peripheral arterial disease. Lancet. 2001 Oct 13;358(9289):1257-64. doi: 10.1016/S0140-6736(01)06351-6. PMID 11675083
- [Background] Meijer WT, Hoes AW, Rutgers D, Bots ML, Hofman A, Grobbee DE. Peripheral arterial disease in the elderly: The Rotterdam Study. Arterioscler Thromb Vasc Biol. 1998 Feb;18(2):185-92. doi: 10.1161/01.atv.18.2.185. PMID 9484982
- [Background] Hirsch AT, Haskal ZJ, Hertzer NR, Bakal CW, Creager MA, Halperin JL, Hiratzka LF, Murphy WR, Olin JW, Puschett JB, Rosenfield KA, Sacks D, Stanley JC, Taylor LM Jr, White CJ, White J, White RA, Antman EM, Smith SC Jr, Adams CD, Anderson JL, Faxon DP, Fuster V, Gibbons RJ, Hunt SA, Jacobs AK, Nishimura R, Ornato JP, Page RL, Riegel B; American Association for Vascular Surgery; Society for Vascular Surgery; Society for Cardiovascular Angiography and Interventions; Society for Vascular Medicine and Biology; Society of Interventional Radiology; ACC/AHA Task Force on Practice Guidelines Writing Committee to Develop Guidelines for the Management of Patients With Peripheral Arterial Disease; American Association of Cardiovascular and Pulmonary Rehabilitation; National Heart, Lung, and Blood Institute; Society for Vascular Nursing; TransAtlantic Inter-Society Consensus; Vascular Disease Foundation. ACC/AHA 2005 Practice Guidelines for the management of patients with peripheral arterial disease (lower extremity, renal, mesenteric, and abdominal aortic): a collaborative report from the American Association for Vascular Surgery/Society for Vascular Surgery, Society for Cardiovascular Angiography and Interventions, Society for Vascular Medicine and Biology, Society of Interventional Radiology, and the ACC/AHA Task Force on Practice Guidelines (Writing Committee to Develop Guidelines for the Management of Patients With Peripheral Arterial Disease): endorsed by the American Association of Cardiovascular and Pulmonary Rehabilitation; National Heart, Lung, and Blood Institute; Society for Vascular Nursing; TransAtlantic Inter-Society Consensus; and Vascular Disease Foundation. Circulation. 2006 Mar 21;113(11):e463-654. doi: 10.1161/CIRCULATIONAHA.106.174526. No abstract available. PMID 16549646
- [Background] Saha SP, Whayne TF Jr, Mukherjee D. Current evidence for antithrombotic therapy after peripheral vascular interventions. Curr Vasc Pharmacol. 2013 Jul;11(4):507-13. doi: 10.2174/1570161111311040014. PMID 22272907
- [Background] Isner JM, Rosenfield K. Redefining the treatment of peripheral artery disease. Role of percutaneous revascularization. Circulation. 1993 Oct;88(4 Pt 1):1534-57. doi: 10.1161/01.cir.88.4.1534. No abstract available. PMID 8403302
- [Background] Andros G. Diagnostic and therapeutic arterial interventions in the ulcerated diabetic foot. Diabetes Metab Res Rev. 2004 May-Jun;20 Suppl 1:S29-33. doi: 10.1002/dmrr.468. PMID 15150810
- [Background] Isner JM, Pieczek A, Schainfeld R, Blair R, Haley L, Asahara T, Rosenfield K, Razvi S, Walsh K, Symes JF. Clinical evidence of angiogenesis after arterial gene transfer of phVEGF165 in patient with ischaemic limb. Lancet. 1996 Aug 10;348(9024):370-4. doi: 10.1016/s0140-6736(96)03361-2. PMID 8709735
- [Background] Baumgartner I, Pieczek A, Manor O, Blair R, Kearney M, Walsh K, Isner JM. Constitutive expression of phVEGF165 after intramuscular gene transfer promotes collateral vessel development in patients with critical limb ischemia. Circulation. 1998 Mar 31;97(12):1114-23. doi: 10.1161/01.cir.97.12.1114. PMID 9537336
- [Background] Kusumanto YH, van Weel V, Mulder NH, Smit AJ, van den Dungen JJ, Hooymans JM, Sluiter WJ, Tio RA, Quax PH, Gans RO, Dullaart RP, Hospers GA. Treatment with intramuscular vascular endothelial growth factor gene compared with placebo for patients with diabetes mellitus and critical limb ischemia: a double-blind randomized trial. Hum Gene Ther. 2006 Jun;17(6):683-91. doi: 10.1089/hum.2006.17.683. PMID 16776576
- [Background] Comerota AJ, Throm RC, Miller KA, Henry T, Chronos N, Laird J, Sequeira R, Kent CK, Bacchetta M, Goldman C, Salenius JP, Schmieder FA, Pilsudski R. Naked plasmid DNA encoding fibroblast growth factor type 1 for the treatment of end-stage unreconstructible lower extremity ischemia: preliminary results of a phase I trial. J Vasc Surg. 2002 May;35(5):930-6. doi: 10.1067/mva.2002.123677. PMID 12021709
- [Background] Isner JM, Walsh K, Symes J, Pieczek A, Takeshita S, Lowry J, Rosenfield K, Weir L, Brogi E, Jurayj D. Arterial gene transfer for therapeutic angiogenesis in patients with peripheral artery disease. Hum Gene Ther. 1996 May 20;7(8):959-88. doi: 10.1089/hum.1996.7.8-959. PMID 8727509
- [Background] Ho HK, Jang JJ, Kaji S, Spektor G, Fong A, Yang P, Hu BS, Schatzman R, Quertermous T, Cooke JP. Developmental endothelial locus-1 (Del-1), a novel angiogenic protein: its role in ischemia. Circulation. 2004 Mar 16;109(10):1314-9. doi: 10.1161/01.CIR.0000118465.36018.2D. Epub 2004 Feb 23. PMID 14981004
- [Background] Rajagopalan S, Mohler ER 3rd, Lederman RJ, Mendelsohn FO, Saucedo JF, Goldman CK, Blebea J, Macko J, Kessler PD, Rasmussen HS, Annex BH. Regional angiogenesis with vascular endothelial growth factor in peripheral arterial disease: a phase II randomized, double-blind, controlled study of adenoviral delivery of vascular endothelial growth factor 121 in patients with disabling intermittent claudication. Circulation. 2003 Oct 21;108(16):1933-8. doi: 10.1161/01.CIR.0000093398.16124.29. Epub 2003 Sep 22. PMID 14504183
- [Background] Creager MA, Olin JW, Belch JJ, Moneta GL, Henry TD, Rajagopalan S, Annex BH, Hiatt WR. Effect of hypoxia-inducible factor-1alpha gene therapy on walking performance in patients with intermittent claudication. Circulation. 2011 Oct 18;124(16):1765-73. doi: 10.1161/CIRCULATIONAHA.110.009407. Epub 2011 Sep 26. PMID 21947297
- [Background] Nikol S, Baumgartner I, Van Belle E, Diehm C, Visona A, Capogrossi MC, Ferreira-Maldent N, Gallino A, Wyatt MG, Wijesinghe LD, Fusari M, Stephan D, Emmerich J, Pompilio G, Vermassen F, Pham E, Grek V, Coleman M, Meyer F; TALISMAN 201 investigators. Therapeutic angiogenesis with intramuscular NV1FGF improves amputation-free survival in patients with critical limb ischemia. Mol Ther. 2008 May;16(5):972-8. doi: 10.1038/mt.2008.33. Epub 2008 Apr 1. PMID 18388929
- [Background] Freedman SB, Isner JM. Therapeutic angiogenesis for coronary artery disease. Ann Intern Med. 2002 Jan 1;136(1):54-71. doi: 10.7326/0003-4819-136-1-200201010-00011. PMID 11777364
- [Background] Novakova V, Sandhu GS, Dragomir-Daescu D, Klabusay M. Apelinergic system in endothelial cells and its role in angiogenesis in myocardial ischemia. Vascul Pharmacol. 2016 Jan;76:1-10. doi: 10.1016/j.vph.2015.08.005. Epub 2015 Aug 5. PMID 26254105
- [Background] Van Raemdonck K, Van den Steen PE, Liekens S, Van Damme J, Struyf S. CXCR3 ligands in disease and therapy. Cytokine Growth Factor Rev. 2015 Jun;26(3):311-27. doi: 10.1016/j.cytogfr.2014.11.009. Epub 2014 Nov 22. PMID 25498524
- [Background] Asahara T, Murohara T, Sullivan A, Silver M, van der Zee R, Li T, Witzenbichler B, Schatteman G, Isner JM. Isolation of putative progenitor endothelial cells for angiogenesis. Science. 1997 Feb 14;275(5302):964-7. doi: 10.1126/science.275.5302.964. PMID 9020076
- [Background] Leeper NJ, Hunter AL, Cooke JP. Stem cell therapy for vascular regeneration: adult, embryonic, and induced pluripotent stem cells. Circulation. 2010 Aug 3;122(5):517-26. doi: 10.1161/CIRCULATIONAHA.109.881441. No abstract available. PMID 20679581
- [Background] Tateishi-Yuyama E, Matsubara H, Murohara T, Ikeda U, Shintani S, Masaki H, Amano K, Kishimoto Y, Yoshimoto K, Akashi H, Shimada K, Iwasaka T, Imaizumi T; Therapeutic Angiogenesis using Cell Transplantation (TACT) Study Investigators. Therapeutic angiogenesis for patients with limb ischaemia by autologous transplantation of bone-marrow cells: a pilot study and a randomised controlled trial. Lancet. 2002 Aug 10;360(9331):427-35. doi: 10.1016/S0140-6736(02)09670-8. PMID 12241713
- [Background] Saigawa T, Kato K, Ozawa T, Toba K, Makiyama Y, Minagawa S, Hashimoto S, Furukawa T, Nakamura Y, Hanawa H, Kodama M, Yoshimura N, Fujiwara H, Namura O, Sogawa M, Hayashi J, Aizawa Y. Clinical application of bone marrow implantation in patients with arteriosclerosis obliterans, and the association between efficacy and the number of implanted bone marrow cells. Circ J. 2004 Dec;68(12):1189-93. doi: 10.1253/circj.68.1189. PMID 15564705
- [Background] Miyamoto K, Nishigami K, Nagaya N, Akutsu K, Chiku M, Kamei M, Soma T, Miyata S, Higashi M, Tanaka R, Nakatani T, Nonogi H, Takeshita S. Unblinded pilot study of autologous transplantation of bone marrow mononuclear cells in patients with thromboangiitis obliterans. Circulation. 2006 Dec 12;114(24):2679-84. doi: 10.1161/CIRCULATIONAHA.106.644203. Epub 2006 Dec 4. PMID 17145986
- [Background] Ruiz-Salmeron R, de la Cuesta-Diaz A, Constantino-Bermejo M, Perez-Camacho I, Marcos-Sanchez F, Hmadcha A, Soria B. Angiographic demonstration of neoangiogenesis after intra-arterial infusion of autologous bone marrow mononuclear cells in diabetic patients with critical limb ischemia. Cell Transplant. 2011;20(10):1629-39. doi: 10.3727/096368910X0177. PMID 22289660
- [Background] Canizo MC, Lozano F, Gonzalez-Porras JR, Barros M, Lopez-Holgado N, Briz E, Sanchez-Guijo FM. Peripheral endothelial progenitor cells (CD133 +) for therapeutic vasculogenesis in a patient with critical limb ischemia. One year follow-up. Cytotherapy. 2007;9(1):99-102. doi: 10.1080/14653240601034708. PMID 17354105
- [Background] Huang P, Li S, Han M, Xiao Z, Yang R, Han ZC. Autologous transplantation of granulocyte colony-stimulating factor-mobilized peripheral blood mononuclear cells improves critical limb ischemia in diabetes. Diabetes Care. 2005 Sep;28(9):2155-60. doi: 10.2337/diacare.28.9.2155. PMID 16123483
- [Background] Lu D, Chen B, Liang Z, Deng W, Jiang Y, Li S, Xu J, Wu Q, Zhang Z, Xie B, Chen S. Comparison of bone marrow mesenchymal stem cells with bone marrow-derived mononuclear cells for treatment of diabetic critical limb ischemia and foot ulcer: a double-blind, randomized, controlled trial. Diabetes Res Clin Pract. 2011 Apr;92(1):26-36. doi: 10.1016/j.diabres.2010.12.010. Epub 2011 Jan 8. PMID 21216483
- [Background] Lasala GP, Silva JA, Minguell JJ. Therapeutic angiogenesis in patients with severe limb ischemia by transplantation of a combination stem cell product. J Thorac Cardiovasc Surg. 2012 Aug;144(2):377-82. doi: 10.1016/j.jtcvs.2011.08.053. Epub 2011 Nov 12. PMID 22079876
- [Background] Hmadcha A, Dominguez-Bendala J, Wakeman J, Arredouani M, Soria B. The immune boundaries for stem cell based therapies: problems and prospective solutions. J Cell Mol Med. 2009 Aug;13(8A):1464-75. doi: 10.1111/j.1582-4934.2009.00837.x. Epub 2009 Jul 6. PMID 19583810
- [Background] Gimble J, Guilak F. Adipose-derived adult stem cells: isolation, characterization, and differentiation potential. Cytotherapy. 2003;5(5):362-9. doi: 10.1080/14653240310003026. PMID 14578098
- [Background] Alvarez Garcia J, Garcia Gomez-Heras S, Riera Del Moral L, Largo C, Garcia-Olmo D, Garcia-Arranz M. The effects of allogenic stem cells in a murine model of hind limb diabetic ischemic tissue. PeerJ. 2017 Aug 21;5:e3664. doi: 10.7717/peerj.3664. eCollection 2017. PMID 28852591
- [Background] Escacena N, Quesada-Hernandez E, Capilla-Gonzalez V, Soria B, Hmadcha A. Bottlenecks in the Efficient Use of Advanced Therapy Medicinal Products Based on Mesenchymal Stromal Cells. Stem Cells Int. 2015;2015:895714. doi: 10.1155/2015/895714. Epub 2015 Jul 27. PMID 26273307
- [Background] Acosta L, Hmadcha A, Escacena N, Perez-Camacho I, de la Cuesta A, Ruiz-Salmeron R, Gauthier BR, Soria B. Adipose mesenchymal stromal cells isolated from type 2 diabetic patients display reduced fibrinolytic activity. Diabetes. 2013 Dec;62(12):4266-9. doi: 10.2337/db13-0896. Epub 2013 Sep 16. PMID 24043757
- [Background] Ramsey SD, Newton K, Blough D, McCulloch DK, Sandhu N, Wagner EH. Patient-level estimates of the cost of complications in diabetes in a managed-care population. Pharmacoeconomics. 1999 Sep;16(3):285-95. doi: 10.2165/00019053-199916030-00005. PMID 10558040
- [Background] Lozano FS, Gonzalez-Porras JR, March JR, Lobos JM, Carrasco E, Ros E. Diabetes mellitus and intermittent claudication: a cross-sectional study of 920 claudicants. Diabetol Metab Syndr. 2014 Feb 17;6(1):21. doi: 10.1186/1758-5996-6-21. PMID 24533798
- [Background] Uccioli L, Meloni M, Izzo V, Giurato L, Merolla S, Gandini R. Critical limb ischemia: current challenges and future prospects. Vasc Health Risk Manag. 2018 Apr 26;14:63-74. doi: 10.2147/VHRM.S125065. eCollection 2018. PMID 29731636
- [Background] Schreuder SM, Hendrix YMGA, Reekers JA, Bipat S. Predictive Parameters for Clinical Outcome in Patients with Critical Limb Ischemia Who Underwent Percutaneous Transluminal Angioplasty (PTA): A Systematic Review. Cardiovasc Intervent Radiol. 2018 Jan;41(1):1-20. doi: 10.1007/s00270-017-1796-9. Epub 2017 Sep 18. PMID 28924874
- [Background] Meloni M, Izzo V, Giurato L, Del Giudice C, Da Ros V, Cervelli V, Gandini R, Uccioli L. Recurrence of Critical Limb Ischemia After Endovascular Intervention in Patients with Diabetic Foot Ulcers. Adv Wound Care (New Rochelle). 2018 Jun 1;7(6):171-176. doi: 10.1089/wound.2017.0778. PMID 29892493
- [Background] Neupane S, Edla S, Maidona E, Sweet MC, Szpunar S, Davis T, LaLonde TA, Mehta RH, Rosman HS, Yamasaki H. Long-term outcomes of patients with diabetes mellitus undergoing percutaneous intervention for popliteal and infrapopliteal peripheral arterial disease. Catheter Cardiovasc Interv. 2018 Jul;92(1):117-123. doi: 10.1002/ccd.27571. Epub 2018 Mar 14. PMID 29536612
- [Background] Spillerova K, Settembre N, Biancari F, Alback A, Venermo M. Angiosome Targeted PTA is More Important in Endovascular Revascularisation than in Surgical Revascularisation: Analysis of 545 Patients with Ischaemic Tissue Lesions. Eur J Vasc Endovasc Surg. 2017 Apr;53(4):567-575. doi: 10.1016/j.ejvs.2017.01.008. Epub 2017 Feb 16. PMID 28215512
- [Derived] Dubsky M, Husakova J, Sojakova D, Fejfarova V, Jude EB. Cell Therapy of Severe Ischemia in People with Diabetic Foot Ulcers-Do We Have Enough Evidence? Mol Diagn Ther. 2023 Nov;27(6):673-683. doi: 10.1007/s40291-023-00667-w. Epub 2023 Sep 22. PMID 37740111
- [Derived] Soria-Juan B, Garcia-Arranz M, Llanos Jimenez L, Aparicio C, Gonzalez A, Mahillo Fernandez I, Riera Del Moral L, Grochowicz L, Andreu EJ, Marin P, Castellanos G, Moraleda JM, Garcia-Hernandez AM, Lozano FS, Sanchez-Guijo F, Villaron EM, Parra ML, Yanez RM, de la Cuesta Diaz A, Tejedo JR, Bedoya FJ, Martin F, Miralles M, Del Rio Sola L, Fernandez-Santos ME, Ligero JM, Morant F, Hernandez-Blasco L, Andreu E, Hmadcha A, Garcia-Olmo D, Soria B. Efficacy and safety of intramuscular administration of allogeneic adipose tissue derived and expanded mesenchymal stromal cells in diabetic patients with critical limb ischemia with no possibility of revascularization: study protocol for a randomized controlled double-blind phase II clinical trial (The NOMA Trial). Trials. 2021 Sep 6;22(1):595. doi: 10.1186/s13063-021-05430-2. PMID 34488845